CLINICAL TRIAL: NCT05589168
Title: 911 Nurse Triage Line Randomized Controlled Trial
Brief Title: 911 Nurse Triage Line
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Lab @ DC (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1-1033362-1
Record Dates: First submitted 2022-10-04; First posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Emergencies
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Triage Nurse (Experimental): Triage nurse
  Interventions: Behavioral: Triage nurse
- No Triage Nurse (Active Comparator): No triage nurse
  Interventions: Behavioral: No triage nurse

INTERVENTIONS:
Behavioral: Triage nurse — Triage nurse joins 911 call
  Arms: Triage Nurse
Behavioral: No triage nurse — Triage nurse does not join 911 call (business as usual)
  Arms: No Triage Nurse

SUMMARY:
Each year, millions of Americans call 911 for time-sensitive issues that don't require Emergency Medical Services (EMS). In need of medical help, these callers may treat 911 as an entry point into the healthcare system, yet an ambulance to the emergency department can harm both their own long-term health and the health of others. In a field experiment in Washington, DC, the investigators randomly assign nurses directly into 911 calls in order to triage low-acuity calls. While other 911 reforms have denied callers access to alternative resources, this effort reforms 911 by offering appropriate care.

ELIGIBILITY:
Inclusion Criteria:

* Low-acuity call

Exclusion Criteria:

* Incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6053 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Ambulance dispatch | During or immediately subsequent to call
  Ambulance is dispatched in response to the 911 call
Ambulance transport | During or immediately subsequent to call
  Caller is transported in dispatched ambulance
ED visit, 24 hours | 24 hours
  Emergency department visit within 24 hours
ED visit, 6 months | 6 months
  Emergency department visit with 6 months
Primary care visit, 24 hours | 24 hours
  Primary care visit within 24 hours
Primary care visit, 6 months | 6 months
  Primary care visit within 6 months
911 use, 24 hours | 24 hours
  Whether caller made subsequent calls to 911 within 24 hours
911 use, 6 months | 6 months
  Whether caller made subsequent calls to 911 within 6 months
Health expenditures | 6 months
  Total dollars and log-transformed dollars of Medicaid health expenditures

CONTACTS AND LOCATIONS:
Locations (1):
- Office of Unified Communications, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Pre-Analysis Plan — https://osf.io/j89ns/